CLINICAL TRIAL: NCT06320288
Title: Analysis of Trunk and Center of Mass Control Development During Gait in Children With Cerebral Palsy
Brief Title: Analysis of Trunk and Center of Mass Control Development During Gait in Children With Cerebral Palsy (VERTEBRAL)
Acronym: VERTEBRAL
Status: Recruiting | Type: Observational
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00505-40
Record Dates: First submitted 2024-02-05; First posted 2024-03-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Children With Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with cerebral palsy: All children will undergo :
  * A neuro-articular assessment
  * A gait analysis on a walking track and with three inertial units to analyze the behavior of their trunk and center of mass during walking.
  * Assessment of gross motor function
  * Static posturography
  * Functional assessment of the trunk
  * Functional assessment of balance
- Children with typical development: All children will undergo :
  * A neuro-articular assessment
  * A gait analysis on a walking track and with three inertial units to analyze the behavior of their trunk and center of mass during walking.
  * Static posturography
  * Functional assessment of the trunk
  * Functional assessment of balance

SUMMARY:
During the acquisition of posturokinetic abilities such as walking, postural control of the trunk is of paramount importance. Indeed, its development is strongly linked to the overall motor function of children. In cerebral palsy (CP), a term that refers to a set of motor disorders following a perinatal lesion, deficits in axial control are present from early childhood. These deficits are strongly correlated with the functional deficits observed in this population. In particular, during walking, deviations of the trunk (amplitudes, accelerations) are observed in the three planes of space. While recent literature increasingly questions the impact of trunk control deficit on the walking of children with CP, elements are still missing for a holistic understanding of the interaction between locomotor and postural disorders in children with CP. In particular, no study has focused on the deviations of trunk control and the center of mass (which is a global indicator of balance strategies) during the development and maturation of walking in children with CP. Therefore, the primary objective of this cross-sectional observational study will be to characterize the development of trunk control and center of mass during walking in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children (< 18 years) with cerebral palsy
* GMFCS I to III
* Independent walking with or without technical walking aids (walker, crutches, etc.)
* Able to understand the instructions of various clinical assessments and functional explorations
* Affiliated with a social security scheme

Exclusion Criteria:

Children with cerebral palsy

* Neuro-orthopaedic surgery of the lower limbs or trunk within the last 12 months
* Botulinum toxin A injections within the last 6 months
* Therapeutic intervention targeting trunk control last 6 months

Typically developing children

* Surgery on lower limbs or trunk last 12 months
* Neurological and/or orthopedic pathology that may influence gait

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with cerebral palsy presenting gait pattern disorders receive consultation and/or care (day or full hospitalization) at the Flavigny-sur-Moselle CMPRE.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Trunk and center-of-mass accelerations and acceleration variability | At the end of the one-day experimental
  In addition to the zeno walking track, inertial computers will be used to record accelerations of the patient's trunk and center of mass as they walk. One will be attached to the sternum, the other to the lumbosacral hinge, using hypoallergenic double-sided tape. A third will be attached to the patient's shoe to synchronize the data from the treadmill and the inertial units. Acceleration variability is calculated in post-processing.

SECONDARY OUTCOMES:
Gait Variability Index | At the beginning of the one-day experimental
  A composite score of gait variability based on spatio-temporal parameters, giving an index of gait regularity. The mean reference score is 100, and a score above 100 indicates that the patient is at least as stable as a patient from a healthy population.
Trunk Control Measurement Scale score (TCMS) | At the beginning of the one-day experimental
  The TCMS scale assesses trunk control in the seated position in three dimensions. The maximum (and best) score is 58 points, of which 20 correspond to static balance, 28 to selective movement control and 10 to the ability to perform dynamic extension movements.
Early Clinical Assessment of Balance score | At the beginning of the one-day experimental
  The Early Clinical Assessment of Balance is an evaluative measure used by clinicians to assess balance in the cerebral palsy population. Scoring is on a 0-100 scale where higher scores equate to better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France